CLINICAL TRIAL: NCT01443104
Title: A Randomized Comparison of a Sirolimus-eluting Stent With Biodegradable Polymer Versus an Everolimus-eluting Stent With a Durable Polymer for Percutaneous Coronary Revascularization
Brief Title: Sirolimus-eluting Stents With Biodegradable Polymer Versus an Everolimus-eluting Stents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Biotronik AG (Industry); University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 065/11
Record Dates: First submitted 2011-09-21; First posted 2011-09-29 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Coronary Artery Disease; Angina Pectoris; Myocardial Infarction
Keywords: coronary artery disease; drug-eluting stents; polymers
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Orsiro Stent (Active Comparator): Sirolimus-eluting Stent with a Biodegradable Polymer
  Interventions: Device: Sirolimus-eluting stent with a bioresorbable polymer (Orsiro)
- Xience Prime Stent (Active Comparator): Everolimus-eluting Stent with a Durable Polymer
  Interventions: Device: Everolimus-eluting stent with a durable polymer

INTERVENTIONS:
Device: Sirolimus-eluting stent with a bioresorbable polymer (Orsiro) — Percutaneous coronary intervention with implantation of a sirolimus-eluting stent with a bioresorbable polymer for coronary artery disease
  Arms: Orsiro Stent
Device: Everolimus-eluting stent with a durable polymer — Percutaneous coronary intervention with implantation of an everolimus-eluting stent with a durable polymer for coronary artery disease
  Arms: Xience Prime Stent

SUMMARY:
Coronary artery stents have improved the safety and efficacy of percutaneous coronary intervention for coronary artery disease. Drug-eluting stents have been shown to decrease neointimal hyperplasia and to reduce the rate of restenosis and target-lesion revascularization as compared to bare-metal stents. Drug-eluting stents consist of a metallic platform and a therapeutic substance that is usually released from a polymer matrix. A previous study utilizing a bioresorbable polymer has demonstrated a favorable safety and efficacy profile in a large-scale clinical trial as compared to a first-generation druf-eluting stent (LEADERS trial).

The objective of the study is to compare the safety and efficacy of a sirolimus-eluting stent with a biodegradable polymer with an everolimus-eluting stent with a durable polymer in a prospective multicenter randomized controlled non-inferiority trial in patients undergoing percutaneous coronary intervention in routine clinical practice.

DETAILED DESCRIPTION:
Background

Coronary artery stents have improved the safety and efficacy of percutaneous coronary interventions compared with balloon angioplasty alone (New Engl J Med 1994; 331:489-495). Notwithstanding, restenosis is still encountered in 20 to 30% of lesions after implantation of bare metal stents (JAMA 2000; 284:1828-36) and may require repeat revascularization procedures with a negative impact on quality of life and health care expenditures. Drug-eluting stents with local, controlled release of therapeutic agents have addressed this problem successfully (Circulation 2003; 107:3003-7). Current drug-eluting stents consist of a metallic stent platform and a therapeutic agent, which is either directly immobilized on the stent surface or released from a polymer matrix. Polymers currently utilized for drug-eluting stents are either biodegradable or non-biodegradable. While biodegradable polymers are released together with the drug and dissolve after a certain period of time, non-biodegradable polymers reside permanently on the stent surface.

First-generation drug-eluting stents utilized sirolimus and paclitaxel for prevention of restenosis. Both drugs are highly lipophilic and show rapid and strong uptake in arterial wall tissue. In addition, Sirolimus (Circulation 2001; 104:852-5) and paclitaxel (Circulation 1997; 96:636-45) have been shown to reduce smooth muscle cell proliferation and neointimal hyperplasia, the principal cause of restenosis after coronary stenting in experimental models. A polymer-encapsulated stent releasing Sirolimus has been compared with the respective bare metal stent in several randomized clinical trials, demonstrating a consistent reduction in angiographic and clinical restenosis (N Engl J Med 2002; 346:1773-80). Similarly, a polymer-based, paclitaxel-eluting stent consistently reduced restenosis and the need for repeated revascularization procedures compared with the respective bare metal stent (N Engl J Med 2004; 350:221-31). A meta-analysis of drug-eluting stent trials confirmed the reduction in restenosis and repeat revascularization procedures for polymer-based, drug-eluting stents (Lancet 2004; 364:583-91). Moreover, the rates of death and myocardial infarction were comparable to those with bare metal stents, attesting to the safety of these devices, which have been approved by the US Food and Drug Administration.

Newer generation drug-eluting stents with durable polymer coating utilize Limus analogues such as everolimus, zotarolimus or novolimus. Everolimus-eluting stents have been compared to first-generation drug-eluting stents in several randomized clinical trials. A pooled analysis of the four largest randomized trials to date comparing everolimus-eluting stents with paclitaxel-eluting stents demonstrated a lower rate of MACE (4.4% versus 7.6%), myocardial infarction (2.1% vs. 4.0%, p<0.001), ischemic TLR (2.3% vs. 4.7%, p<0.001), and definite stent thrombosis (0.4% vs. 1.2%, p<0.001) in favor of EES, whereas there was no difference with regard to overall and cardiac mortality (Stone GW. The XIENCE V - PROMUS Everolimus-Eluting Stent: New Insights from the SPIRIT/COMPARE Meta-analysis and other randomized trials. Presentation at Transcatheter Cardiovascular Therapeutics, September 22nd 2010). At the same time several trials comparing everolimus-eluting stents with sirolimus-eluting stents reported favorable performance of everolimus-eluting stents. In a randomized trial enrolling 2'774 patients everolimus-eluting stents were non-inferior compared with sirolimus-eluting stents at nine months with regard to MACE (4.9% vs. 5.2%, HR 0.94, 0.67-1.31) and TLR (1.4% vs. 1.7%, HR 0.87, 0.48-1.58) (N Engl J Med 2010;362(28):1663-74). Likewise, event rates at two years were similar for everolimus-eluting stents and sirolimus-eluting stents (3.7% versus 4.3%, p=0.85) in a randomized controlled trial comparing EES, SES, and BMS in large vessels (stent diameter >3.0 mm), whereas TVR was lower with both EES (3.7%) and SES (4.3%) as compared with bare-metal stents (10.3%, P=0.005 vs SES, P=0.002 vs EES) (N Engl J Med 2010;363(24):2310-9). A propensity-score matched comparison of EES and SES reported lower event rates of myocardial infarction (3.3% versus 5.0%, HR 0.62, 95% CI 0.42-0.92, P=0.017) in part due to a lower risk of stent thrombosis (definite or probable 2.5% versus 4.0%, HR 0.64, 95% CI 0.41-0.98, P=0.041), as well as a lower rate of target vessel revascularization (7.0% versus 9.6%, HR 0.75, 95% CI 0.57-0.99, P=0.039) for EES at three years while mortality was similar (Windecker S. Long-term comparison of Everolimus-eluting and Sirolimus-eluting Stents for coronary revascularization 1 (LESSON1) study. Presentation at the European Society of Cardiology meeting, Stockholm, Sweden, 31st August 2010. 2010).

A previous study utilizing a bioresorbable polymer has demonstrated a favorable safety and efficacy profile in a large-scale clinical trial as compared to a first-generation drug-eluting stent. Among 1,707 patients randomized to either a biolimus-eluting stent with a bioresorbable polymer or a sirolimus-eluting stent with a durable polymer no significant differences with regard to the primary endpoint of cardiac death, myocardial infarction or target-vessel revascularization were observed (9.2% versus 10.5%, HR 0.88, 95% CI 0.64-1.19;: p=0.39)(Lancet 2008;372:1163-73.)

Objective

The objective of the study is to compare the safety and efficacy of a sirolimus-eluting stent with a biodegradable polymer with an everolimus-eluting stent with a durable polymer in a prospective multicenter randomized controlled non-inferiority trial in patients undergoing percutaneous coronary intervention in routine clinical practice.

Methods

Design: Prospective, multi-center, randomized, non-inferiority trial. Patients will be randomized in a single-blind fashion (1:1 randomization) to either the Orsiro® Stent system (Sirolimus-eluting stent with a biodegradable polymer) with the Xience PRIME® stent system (Everolimus-eluting stent with a durable polymer).

Primary endpoint: Target lesion failure (TLF), defined as the composite of cardiac death, target vessel myocardial infarction (MI), and clinically driven target-lesion revascularization (TLR).

Inclusion Criteria: "Real world, all comer" patients with symptomatic coronary artery disease including patients with chronic stable angina, silent ischemia, and acute coronary syndromes including NSTE-ACS and STE-ACS, and presence of one or more coronary artery stenoses >50% in a native coronary artery or a saphenous bypass graft which can be treated with a stent ranging in diameter from 2.25 to 4.0 mm and can be covered with one or multiple stents.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Symptomatic coronary artery disease including patients with chronic stable angina, silent ischemia, and acute coronary syndromes including NSTE-ACS and STE-ACS
* Presence of one or more coronary artery stenoses >50% in a native coronary artery or a saphenous bypass graft which can be treated with a stent ranging in diameter from 2.25 to 4.0 mm and can be covered with one or multiple stents
* No limitation on the number of treated lesions, and vessels, and lesion length

Exclusion Criteria

* Pregnancy
* Known intolerance to aspirin, clopidogrel, heparin, stainless steel, Sirolimus, Everolimus or contrast material
* Inability to provide informed consent
* Currently participating in another trial before reaching first endpoint
* Planned surgery within 6 months of PCI unless dual antiplatelet therapy is maintained throughout the peri-surgical period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2119 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Target lesion failure (TLF), defined as the composite of cardiac death, target vessel Q-wave or non-Q wave myocardial infarction (MI), and clinically driven target lesion revascularization (TLR) and emergent coronary artery bypass grafting (CABG) | 12 months

SECONDARY OUTCOMES:
Number of patients with target lesion revascularization (TLR) | 30 days
Number of patients with target lesion revascularization (TLR) | 1 year
Number of patients with target lesion revascularization (TLR) | 2 years
Number of patients with target lesion revascularization (TLR) | 5 years
Clinically indicated and not clinically indicated target vessel revascularization (TVR) | 30 days
Clinically indicated and not clinically indicated target vessel revascularization (TVR) | 1 year
Clinically indicated and not clinically indicated target vessel revascularization (TVR) | 2 years
Clinically indicated and not clinically indicated target vessel revascularization (TVR) | 5 years
TLF composite of cardiac death, target vessel Q-wave or non-Q wave myocardial infarction (MI) | 30 days
TLF composite of cardiac death, target vessel Q-wave or non-Q wave myocardial infarction (MI) | 2 years
TLF composite of cardiac death, target vessel Q-wave or non-Q wave myocardial infarction (MI) | 5 years
All-cause mortality | 30 days
All-cause mortality | 1 year
All-cause mortality | 2 years
All-cause mortality | 5 years
Definite stent thrombosis | 30 days
Definite stent thrombosis | 1 year
Definite stent thrombosis | 2 years
Definite stent thrombosis | 3 years
Definite stent thrombosis | 5 years
Myocardial infarction (Q-wave and NQWMI) | 30 days
Myocardial infarction (Q-wave and NQWMI) | 1 year
Myocardial infarction (Q-wave and NQWMI) | 2 years
Myocardial infarction (Q-wave and NQWMI) | 3 years
Myocardial infarction (Q-wave and NQWMI) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Windecker, Principal Investigator — Department of Cardiology, Bern University Hospital, Switzerland
Locations (9):
- Switzerland (9):
  - Kantonsspital Aarau, Aarau
  - Universitätsklinik Basel, Basel
  - Department of Cardiology, Bern University Hospital, Bern
  - HFR Freiburg, Fribourg
  - Hôpitaux Universitaires de Genève, Geneva
  - Service de cardiologie CHUV, Lausanne
  - Luzerner Kantonsspital, Lucerne
  - Kantonsspital St. Gallen, Sankt Gallen
  - Stadtspital Triemli, Zurich

REFERENCES:
- [Result] Zbinden R, Piccolo R, Heg D, Roffi M, Kurz DJ, Muller O, Vuilliomenet A, Cook S, Weilenmann D, Kaiser C, Jamshidi P, Franzone A, Eberli F, Juni P, Windecker S, Pilgrim T. Ultrathin Strut Biodegradable Polymer Sirolimus-Eluting Stent Versus Durable-Polymer Everolimus-Eluting Stent for Percutaneous Coronary Revascularization: 2-Year Results of the BIOSCIENCE Trial. J Am Heart Assoc. 2016 Mar 15;5(3):e003255. doi: 10.1161/JAHA.116.003255. PMID 26979080
- [Result] Franzone A, Pilgrim T, Heg D, Roffi M, Tuller D, Vuilliomenet A, Muller O, Cook S, Weilenmann D, Kaiser C, Jamshidi P, Raber L, Stortecky S, Wenaweser P, Juni P, Windecker S. Clinical outcomes according to diabetic status in patients treated with biodegradable polymer sirolimus-eluting stents versus durable polymer everolimus-eluting stents: prespecified subgroup analysis of the BIOSCIENCE trial. Circ Cardiovasc Interv. 2015 Jun;8(6):e002319. doi: 10.1161/CIRCINTERVENTIONS.114.002319. PMID 26043895
- [Result] Pilgrim T, Piccolo R, Heg D, Roffi M, Tuller D, Vuilliomenet A, Muller O, Cook S, Weilenmann D, Kaiser C, Jamshidi P, Khattab AA, Taniwaki M, Rigamonti F, Nietlispach F, Blochlinger S, Wenaweser P, Juni P, Windecker S. Biodegradable polymer sirolimus-eluting stents versus durable polymer everolimus-eluting stents for primary percutaneous coronary revascularisation of acute myocardial infarction. EuroIntervention. 2016 Dec 10;12(11):e1343-e1354. doi: 10.4244/EIJY15M12_09. PMID 26690319
- [Result] Pilgrim T, Heg D, Roffi M, Tuller D, Muller O, Vuilliomenet A, Cook S, Weilenmann D, Kaiser C, Jamshidi P, Fahrni T, Moschovitis A, Noble S, Eberli FR, Wenaweser P, Juni P, Windecker S. Ultrathin strut biodegradable polymer sirolimus-eluting stent versus durable polymer everolimus-eluting stent for percutaneous coronary revascularisation (BIOSCIENCE): a randomised, single-blind, non-inferiority trial. Lancet. 2014 Dec 13;384(9960):2111-22. doi: 10.1016/S0140-6736(14)61038-2. Epub 2014 Sep 1. PMID 25189359
- [Result] Pilgrim T, Piccolo R, Heg D, Roffi M, Tuller D, Muller O, Moarof I, Siontis GCM, Cook S, Weilenmann D, Kaiser C, Cuculi F, Hunziker L, Eberli FR, Juni P, Windecker S. Ultrathin-strut, biodegradable-polymer, sirolimus-eluting stents versus thin-strut, durable-polymer, everolimus-eluting stents for percutaneous coronary revascularisation: 5-year outcomes of the BIOSCIENCE randomised trial. Lancet. 2018 Sep 1;392(10149):737-746. doi: 10.1016/S0140-6736(18)31715-X. Epub 2018 Aug 28. PMID 30170848
- [Derived] Haner JD, Rohla M, Losdat S, Iglesias JF, Muller O, Eeckhout E, Kurz D, Weilenmann D, Kaiser C, Tapponnier M, Roffi M, Heg D, Windecker S, Pilgrim T. Ultrathin-strut vs thin-strut drug-eluting stents for multi and single-stent lesions: A lesion-level subgroup analysis of 2 randomized trials. Am Heart J. 2023 Sep;263:73-84. doi: 10.1016/j.ahj.2023.05.004. Epub 2023 May 14. PMID 37192697
- [Derived] Iglesias JF, Muller O, Losdat S, Roffi M, Kurz DJ, Weilenmann D, Kaiser C, Heg D, Windecker S, Pilgrim T. Complex primary percutaneous coronary intervention with ultrathin-strut biodegradable versus thin-strut durable polymer drug-eluting stents in patients with ST-segment elevation myocardial infarction: A subgroup analysis from the BIOSTEMI randomized trial. Catheter Cardiovasc Interv. 2023 Mar;101(4):687-700. doi: 10.1002/ccd.30600. Epub 2023 Feb 19. PMID 36807456
- [Derived] Iglesias JF, Heg D, Roffi M, Degrauwe S, Tuller D, Muller O, Brinkert M, Cook S, Weilenmann D, Kaiser C, Cuculi F, Valgimigli M, Juni P, Windecker S, Pilgrim T. Five-Year Outcomes With Biodegradable-Polymer Sirolimus-Eluting Stents Versus Durable-Polymer Everolimus-Eluting Stents in Patients With Acute Coronary Syndrome: A Subgroup Analysis of the BIOSCIENCE Trial. Cardiovasc Revasc Med. 2022 Jan;34:3-10. doi: 10.1016/j.carrev.2021.02.008. Epub 2021 Feb 25. PMID 33653633
- [Derived] Iglesias JF, Heg D, Roffi M, Tuller D, Lanz J, Rigamonti F, Muller O, Moarof I, Cook S, Weilenmann D, Kaiser C, Cuculi F, Valgimigli M, Juni P, Windecker S, Pilgrim T. Five-Year Outcomes in Patients With Diabetes Mellitus Treated With Biodegradable Polymer Sirolimus-Eluting Stents Versus Durable Polymer Everolimus-Eluting Stents. J Am Heart Assoc. 2019 Nov 19;8(22):e013607. doi: 10.1161/JAHA.119.013607. Epub 2019 Nov 7. PMID 31696762
- [Derived] Iglesias JF, Heg D, Roffi M, Tuller D, Noble S, Muller O, Moarof I, Cook S, Weilenmann D, Kaiser C, Cuculi F, Haner J, Juni P, Windecker S, Pilgrim T. Long-Term Effect of Ultrathin-Strut Versus Thin-Strut Drug-Eluting Stents in Patients With Small Vessel Coronary Artery Disease Undergoing Percutaneous Coronary Intervention: A Subgroup Analysis of the BIOSCIENCE Randomized Trial. Circ Cardiovasc Interv. 2019 Aug;12(8):e008024. doi: 10.1161/CIRCINTERVENTIONS.119.008024. Epub 2019 Aug 6. PMID 31525083
- [Derived] Koskinas KC, Siontis GC, Piccolo R, Franzone A, Haynes A, Rat-Wirtzler J, Silber S, Serruys PW, Pilgrim T, Raber L, Heg D, Juni P, Windecker S. Impact of Diabetic Status on Outcomes After Revascularization With Drug-Eluting Stents in Relation to Coronary Artery Disease Complexity: Patient-Level Pooled Analysis of 6081 Patients. Circ Cardiovasc Interv. 2016 Feb;9(2):e003255. doi: 10.1161/CIRCINTERVENTIONS.115.003255. PMID 26823484
- [Derived] Campos CM, Costa F, Garcia-Garcia HM, Bourantas C, Suwannasom P, Valgimigli M, Morel MA, Windecker S, Serruys PW. Anatomic characteristics and clinical implications of angiographic coronary thrombus: insights from a patient-level pooled analysis of SYNTAX, RESOLUTE, and LEADERS Trials. Circ Cardiovasc Interv. 2015 Apr;8(4):e002279. doi: 10.1161/CIRCINTERVENTIONS.114.002279. PMID 25825008
- [Derived] Pilgrim T, Roffi M, Tuller D, Muller O, Vuilliomenet A, Cook S, Weilenmann D, Kaiser C, Jamshidi P, Heg D, Juni P, Windecker S. Randomized comparison of biodegradable polymer sirolimus-eluting stents versus durable polymer everolimus-eluting stents for percutaneous coronary revascularization: rationale and design of the BIOSCIENCE trial. Am Heart J. 2014 Sep;168(3):256-61. doi: 10.1016/j.ahj.2014.06.004. Epub 2014 Jun 6. PMID 25173535